CLINICAL TRIAL: NCT04857827
Title: A Randomized Active-controlled Study to Evaluate Safety and Tolerability of QLS-101 Versus Timolol Preservative Free (PF) Ophthalmic Solution in Subjects With Normal Tension Glaucoma (NTG)
Brief Title: A Study to Evaluate Safety and Tolerability of QLS-101 in NTG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qlaris Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QC-202
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Normal Tension Glaucoma (NTG)
Keywords: low tension glaucoma (LTG); glaucoma
MeSH Terms: conditions — Low Tension Glaucoma; Glaucoma | interventions — Ophthalmic Solutions; Timolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Study subjects, Investigators and their staff, and Sponsor personnel involved with the conduct and monitoring of the study will be masked to the investigational product (IP) identity until after the final database is locked. IPs will be provided in identical-appearing pouches to maintain masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- QLS-101 ophthalmic solution 1.0% (Experimental): Ophthalmic solution once daily (QD) dosing in both eyes (OU) for 14 days followed by 14 days of twice daily (BID) dosing.
  Interventions: Drug: QLS-101
- Timolol maleate PF 0.5% ophthalmic solution (Active Comparator): Ophthalmic solution QD OU dosing for 14 days followed by 14 days BID OU dosing.
  Interventions: Drug: Timolol maleate PF 0.5% ophthalmic solution
- QLS-101 ophthalmic solution 2.0% (Experimental): Ophthalmic solution QD OU dosing for 14 days followed by 14 days BID OU dosing.
  Interventions: Drug: QLS-101

INTERVENTIONS:
Drug: QLS-101 — Ophthalmic solution QD OU dosing for 14 days followed by 14 days BID OU dosing.
  Other Names: QLS-101 ophthalmic solution
  Arms: QLS-101 ophthalmic solution 1.0%; QLS-101 ophthalmic solution 2.0%
Drug: Timolol maleate PF 0.5% ophthalmic solution — Ophthalmic solution QD OU dosing for 14 days followed by 14 days BID OU dosing.
  Other Names: Timolol
  Arms: Timolol maleate PF 0.5% ophthalmic solution

SUMMARY:
A randomized active-controlled multi-site double-masked 28 day study to evaluate the safety and tolerability of QLS-101 versus timolol maleate Preservative Free (PF) 0.5% ophthalmic solution in subjects with normal tension glaucoma

ELIGIBILITY:
Inclusion Criteria:

1. Visual acuity +1.0 logMAR or better
2. Willing to give informed consent
3. Ability to washout from current intraocular pressure lowering medications -

Exclusion Criteria:

1. All secondary glaucomas
2. Previous glaucoma intraocular or laser surgery (selective laser trabeculoplasty permitted when done 18 months or longer from Screening)
3. Refractive surgery
4. Ocular infection or inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Ocular safety | 86 days
  Number of participants with treatment-related adverse events will be monitored

SECONDARY OUTCOMES:
Ocular hypotensive efficacy | 14 days
  Number of participants with intraocular pressure reduction from baseline will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: B. Wirostko, M.D., Study Director — Qlaris Bio, Inc.
Locations (1):
- Vance Thompson Vision, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: company website — https://qlaris.bio